CLINICAL TRIAL: NCT05758480
Title: Characterization of the Immunometabolic Signature in Long COVID-19.
Acronym: LoCo-ImMet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LoCo-ImMet
Record Dates: First submitted 2023-03-01; First posted 2023-03-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Long COVID
Keywords: Long COVID; immunometabolic; immunometabolic signatures
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Two groups:
  1. Patients with Long COVID
  2. Control group composed of patients who recovered from COVID-19 without persistent symptoms.
  Each patient with Long COVID is paired with a matched control, based on age, sex, and date of COVID-19.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Long COVID (Experimental)
  Interventions: Biological: Blood sample (at inclusion and 6 months later); Other: Patient questionnaires (at inclusion and 6 months later)
- COVID-19 recovered patients (Control) (Active Comparator)
  Interventions: Biological: Blood sample (at inclusion and 6 months later); Other: Patient questionnaires (at inclusion and 6 months later)

INTERVENTIONS:
Biological: Blood sample (at inclusion and 6 months later) — (56ml of blood, 8 tubes) 3 heparin, 1 EDTA , 2 SST, 2 CPT
Other: Patient questionnaires (at inclusion and 6 months later) — (4 questionnaires) Symptoms in the last week, Fatigue Impact Scale (FIS), Short-Form 36 (SF-36) and Nijmegen.

SUMMARY:
The primary objective of this study is to identify immunometabolic signatures associated with Long COVID in plasma and peripheral blood mononuclear cells (PBMC).

DETAILED DESCRIPTION:
The mechanisms underlying Long COVID remain poorly understood. Among the symptoms most frequently reported by patients with long COVID, some (fatigue, neurocognitive disorders, muscular weakness) are similar to those reported by patients with innate or acquired abnormalities in energy metabolism, suggesting that metabolic changes could play a role in the disease. On the other hand, other studies have shown that COVID-19 induces an immune dysregulation that could persist after recovery.

The hypothesis of this study is that there are subtle but detectable immunometabolic changes in plasma and PBMC of patients with long COVID. The identification of these specific signatures would help to better understand the physiopathology of this disease and to identify possible therapeutic strategies .

The primary objective of this study is to identify immunometabolic signatures in plasma and peripheral blood mononuclear cells (PBMC) of patients with long COVID, as compared to patients who recovered from COVID-19 without prolonged symptoms.

ELIGIBILITY:
A/ Inclusion Criteria:

* For all patients:

  * Age > 18 years
  * Symptomatic COVID-19 diagnosed after 01JAN2021, confirmed by RT-PCR or Antigen test
  * Last SARS-CoV-2 infection diagnosed more than 12 weeks before inclusion
  * Patient covered by the French health insurance
  * Signature of the informed consent
* For patient with Long COVID :

  * At least one of the following symptoms during the week preceding inclusion: abnormal fatigue, dyspnoea sine materia, abnormal pain (chest, joint, muscle, headache), unusual neurocognitive disorders (concentration disorders, "brain fog", language/memory disorders, paraesthesia)
  * Absence of Return to Usual Health after SARS-CoV-2 infection (patient declaration)
  * Absence of alternative diagnosis for the symptoms
* For COVID-19 recovered patient (Control) :

  * None of the following symptoms in the 3 week before inclusion: abnormal fatigue, dyspnoea sine materia, abnormal pain (chest, joint, muscle, headache), unusual neurocognitive disorders (concentration disorders, "brain fog", language/memory disorders, paraesthesia)
  * Return to Usual Health after SARS-CoV-2 infection (patient declaration)

B/ Exclusion Criteria:

* History of severe COVID-19 (Hospitalization)
* Symptoms caused by sequelae of SARS-CoV-2 infection (in particular, persistence of lung parenchymal abnormalities : pulmonary fibrosis, persistent alveolitis on CT-Scan)
* Significant Depression or anxiety symptoms, as assessed by a > 10 score on the A or D items of the Hospital anxiety and depression scale (HAD)
* Presence of one of the following diseases:

  * Inborn errors of metabolism
  * estimated Glomerular filtration rate < 30 ml/min (MDRD)
  * Autoimmune disease
  * Immunosuppressive treatment or immune deficiency
  * Symptomatic heart failure
  * Respiratory failure (COPD stage ≥ 3 or oxygen therapy)
  * Solid cancer or active blood disease
  * Severe malnutrition (albumin < 30 g/L or weight loss ≥10% in 6 months)
  * Obesity with BMI ≥ 35 kg/m²
  * Diabetes not controlled by diet alone
* Pregnant, breastfeeding or parturient women
* Deprivation of liberty by judicial or administrative decision
* Mandatory Psychiatric Care
* Protected by decision of law
* Unable to express consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Presence of immunometabolic signatures specific of Long COVID in the plasma and mononuclear cells | 18 months
  Statistical analyzes (multivariate) by Orthogonal Projections to Latent Structures Discriminant Analysis (OPLS-DA) (Q2Ycum > 0.5, P-value (CV-ANOVA) ≤0.05, Q2Ycum, test permutations <0) or the median (AUROC test sets) ≥ 0.8 and the median of the p-values associated with the AUROCs of the test sets ≤ 0.05 in the plasma and/or the PBMCs.
Concentration of metabolites and immune mediators in the plasma and mononuclear cells | 18 months
  Comparison of metabolites and immune mediators in the blood and PBMC of patients with long COVID will be compared with those of control patients using statistical tests after correction of the alpha risk.

SECONDARY OUTCOMES:
Changes in immuno-metabolic signatures 6 months after the initial assessment | 18 months
  Significant changes in concentration of metabolites and immune mediators 6 month after inclusion, in comparison with the initial assessment, will be identifed using paired statistical tests with correction of the alpha risk
Proportion of patients with clinical improvement (return to normal life) at 6 months with correction of the immuno-metabolic signature | 18 months
  The correlation between clinical signs of long COVID and the immuno-metabolic signature specific of long COVID identified in the study will be assessed 6 months after inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent DUBEE, MD, PhD, Principal Investigator — Angers University Hospital; Valérie DUBUS, MD, Principal Investigator — Angers University Hospital
Locations (1):
- Angers University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request. Only de-identified data will be shared. Any data collected during the study may be shared. The protocol will be shared initially. Other documents may be shared at a later date upon request (e.g., the CRF to allow a collaborator to select the data they wish to access). The recipients of the data will be researchers. The data will be available for any purpose deemed relevant by the study investigator, based on a protocol provided by the requester, after verification of the obtaining of regulatory approvals, including the favorable opinion of an ethics committee.
Supporting Information: Study Protocol
Time Frame: The data will be shared after signing a negotiated data transfer agreement ( data access agreement), for the duration specified in the agreement.
Access Criteria: The data will be made available via secure transfer (sharing platform approved by the university hospital: BlueFiles or Oodrive).